CLINICAL TRIAL: NCT02132299
Title: Phase 1, Dose Escalation, Randomized Controlled Trial to Evaluate the Safety, Immunogenicity and Efficacy of Intravenously Administered Attenuated Plasmodium Falciparum Sporozoite Vaccine (PfSPZ Vaccine) in Tanzanian Adults
Brief Title: Dose Escalation, Randomized Controlled Trial to Evaluate the Safety, Immunogenicity and Efficacy of Intravenously Administered Attenuated Plasmodium Falciparum Sporozoite Vaccine (PfSPZ Vaccine) in Tanzanian Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Ifakara Health Institute (Other); Swiss Tropical & Public Health Institute (Other); Tanzania Commission for Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BSPZV1
Record Dates: First submitted 2014-04-29; First posted 2014-05-07 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Malaria; Plasmodium Falciparum Malaria
Keywords: Malaria; Plasmodium falciparum malaria; PfSPZ Vaccine; PfSPZ Challenge; Controlled human malaria infection (CHMI)
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group 1 (Experimental): Three volunteers will receive 3 ascending doses of PfSPZ Vaccine by IV administration four weeks apart. The three doses are 3x10^4, 1.35x10^5, and 2.7x10^5 PfSPZ. This is the safety group that will be inoculated first before all others for demonstration of safety and will be followed up for assessment of safety after the completion of the three doses. The follow up will be at weeks 1, 2, 4, 8 and 24 after completion of vaccination. Volunteers in Group 1 will not undergo CHMI. Group 1 is unblinded.
  Interventions: Biological: PfSPZ Vaccine
- Group 2(A) (Experimental): Group 2: Two sub groups: 2A and 2B. Grp 2A (n=20) receives 5 vaccinations IV of 1.35x10^5 PfSPZ Vaccine; 4 doses at 4 wk intervals; 5th dose at 8 wks after 4th dose. Grp 2 starts 1 wk after Grp 1 has completed 2nd dose; and received clearance from Safety Monitoring Committee (SMC). Grp 2 starts with 4 volunteers (3 safety + 1 placebo control to maintain blinding) receiving their first doses (at each dosing time point) before the remaining 20 volunteers in Grp 2. The remaining 20 volunteers start inoculations 48 hrs after first 4 safety volunteers at each dosing time point. Three weeks after last immunization, Grp 2 will undergo the first CHMI by IV injection of 3.2x10^3 PfSPZ Challenge (NF54). 24 weeks after the last immunization, volunteers from Grp 2 who underwent the first CHMI and did not become infected will have a second CHMI by IV injection of 3.2x10^3 PfSPZ Challenge (NF54).
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge
- Group 2(B) (Placebo Comparator): Group 2: Two sub groups: 2A and 2B. Grp 2B (n=4) receives 5 placebo injections of normal saline (NS) by IV administration; 4 doses at 4 wk intervals; 5th dose at 8 wks after 4th dose. Grp 2 starts 1 wk after Grp 1 has completed 2nd dose; and received clearance from Safety Monitoring Committee (SMC). Grp 2 starts with 4 volunteers (3 safety + 1 placebo control to maintain blinding) receiving their first doses (at each dosing time point) before the remaining 20 volunteers in Grp 2. The remaining 20 volunteers start inoculations 48 hrs after first 4 safety volunteers at each dosing time point. Three weeks after last placebo injection, Grp 2 will undergo the first CHMI by IV injection of 3.2x10^3 PfSPZ Challenge (NF54).
  Interventions: Biological: Normal Saline (Placebo); Biological: PfSPZ Challenge
- Group 3(A) (Experimental): Group 3: Two sub groups: 3A and 3B. Grp 3A (n=20) receives 5 vaccinations IV of 2.7x10^5 PfSPZ Vaccine; 4 doses at 4 wk intervals; 5th dose at 8 wks after 4th dose. Grp 3 starts 1 wk after Grp 1 has completed 3rd dose; and received clearance from Safety Monitoring Committee (SMC). Grp 3 starts with 4 volunteers (3 safety + 1 placebo control to maintain blinding) receiving their first doses (at each dosing time point) before the remaining 20 volunteers in Grp 3. The remaining 20 volunteers start inoculations 48 hrs after first 4 safety volunteers at each dosing time point. Three weeks after last immunization, Grp 3 will undergo the first CHMI by IV injection of 3.2x10^3 PfSPZ Challenge (NF54). 24 weeks after the last immunization, volunteers from Grp 3 who underwent the first CHMI and did not become infected will have a second CHMI by IV injection of 3.2x10^3 PfSPZ Challenge (NF54).
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge
- Group 3(B) (Placebo Comparator): Group 3: Two sub groups: 3A and 3B. Grp 3B (n=4) receives 5 placebo injections of normal saline (NS) by IV administration; 4 doses at 4 wk intervals; 5th dose at 8 wks after 4th dose. Grp 3 starts 1 wk after Grp 1 has completed 3rd dose; and received clearance from Safety Monitoring Committee (SMC). Grp 3 starts with 4 volunteers (3 safety + 1 placebo control to maintain blinding) receiving their first doses (at each dosing time point) before the remaining 20 volunteers in Grp 3. The remaining 20 volunteers start inoculations 48 hrs after first 4 safety volunteers at each dosing time point. Three weeks after last placebo injection, Grp 3 will undergo the first CHMI by IV injection of 3.2x10^3 PfSPZ Challenge (NF54).
  Interventions: Biological: Normal Saline (Placebo); Biological: PfSPZ Challenge
- Group 4 (Experimental): The fourth group will include 6 volunteers who will be unblinded and will receive 5 vaccinations of 2.7 x 10^5 PfSPZ Vaccine by IV administration. Four vaccinations at 4 weeks intervals of 2.7x10^5 PfSPZ will be given and the fifth dose will be administered 8 weeks after the 4th. Volunteers from Group 4 will start their vaccinations 48 hours after the four safety volunteers from Group 3 have received their first dose, at each dosing time point. This group will participate in only one CHMI assessment at 24 weeks to assess duration of protection at 24 weeks.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge
- Group 5 (Placebo Comparator): The 5th group will be divided into 3 sub groups 5A, 5B, 5C, who will be screened and recruited to serve as unblinded controls for the 1st and 2nd CHMI at 3 and 24 weeks. They will participate only in the screening and 4 weeks follow up of the 1st and 2nd CHMI assessments. Group 5A (n=2) will be challenged at the time of the 3-week CHMI of Group 2. Group 5B (n=2) will be challenged at the time of the 3-week CHMI of Group 3. Groups 5A and 5B will supplement the 4 NS- injected volunteers as infectivity controls, totaling 6 altogether. Group 5C (n=6) will be challenged at the time of the 24-week CHMI for Groups 3 and 4.
  Interventions: Biological: PfSPZ Challenge

INTERVENTIONS:
Biological: PfSPZ Vaccine — Aseptic, purified, vialed, metabolically active, non-replicating (live, radiation attenuated) cryopreserved Plasmodium falciparum sporozoites (PfSPZ)
  Arms: Group 1; Group 2(A); Group 3(A); Group 4
Biological: Normal Saline (Placebo)
  Arms: Group 2(B); Group 3(B)
Biological: PfSPZ Challenge — Live, infectious, aseptic, purified, vialed, cryopreserved Plasmodium falciparum sporozoites (PfSPZ) for CHMI
  Arms: Group 2(A); Group 2(B); Group 3(A); Group 3(B); Group 4; Group 5

SUMMARY:
This trial will evaluate whether relatively non-immune populations in endemic countries can effectively generate significant cellular and humoral immune responses that confer protection against P. falciparum infection after inoculation of aseptic, purified, vialed, metabolically active, non-replicating (live, radiation attenuated) Plasmodium falciparum sporozoites (PfSPZ Vaccine) administered intravenously (IV).

DETAILED DESCRIPTION:
This is a single center, Phase 1, dose escalating, randomized, double blind, controlled trial. Seventy-three healthy male volunteers, aged 18 to 35 years will be recruited. The study will have 5 study groups that will include 49 volunteers who will be intravenously injected with PfSPZ Vaccine, 8 control volunteers who will receive normal saline and 16 additional control volunteers who will be recruited at the time of controlled human malaria infection (CHMI) at 3 and 24 weeks. The control volunteers will help better assess the occurrence of AEs compared to background disease patterns that occur in this tropical area, and the performance of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged between 18 - 35 years.
* Good health status based on history and clinical examination.
* Long term or permanent resident in or near Dar-es-Salaam.
* Able and willing to complete the study visit schedule over the one year follow up period, including the hospitalizations required for protocol compliance.
* Able and willing to complete the informed consent process conducted in English.
* Demonstrate understanding of the study and procedures by answering 20 questions from the Protocol & Study Procedures Understanding Checklist correctly with a maximum of two attempts.
* Agrees to inform study doctor of medical conditions and contraindications for participation in the study.
* Agrees to provide contact information to the study team for a household member who will serve as an emergency contact during trial participation.
* Willing to be attended by a study doctor and take medications, which may be prescribed by a study doctor, during study participation.
* Reachable (24/7) by mobile phone during the whole study period.
* Agrees not to participate in another study during the study period.
* Agrees not to donate blood during the study period.
* Willing to undergo HIV, hepatitis B and hepatitis C testing.
* Willing to undergo controlled human malaria infection (CHMI).

Exclusion Criteria:

* History of malaria in the past 5 years.
* Positive for malaria by thick blood smear at screening.
* Plans to travel outside the Dar-es-Salaam or Coast Region in first 12 months of the study.
* Previous receipt of an investigational malaria vaccine.
* Antibodies to parasites or selected parasite protein(s) above acceptable cut off established for the site
* History of arrhythmias or prolonged QT-interval or other cardiac disease or clinically significant abnormalities in electrocardiogram (ECG) at screening.
* History or indication of a history of drug or alcohol abuse interfering with normal social function.
* Use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months of study enrollment (inhaled and topical corticosteroids are allowed).
* Ongoing condition that could interfere with the interpretation of the study results or compromise the health of the volunteer.
* History of diabetes mellitus or cancer.
* Body Mass Index (BMI) below 18 or above 30 kg/m2.
* Any clinically significant deviation from the normal range in biochemistry or hematology blood tests or in urine analysis or electrolytes.
* Positive HIV, Hepatitis B virus or Hepatitis C virus tests.
* Participation in any other clinical study within 30 days prior to study enrollment.
* Known hypersensitivity, allergy, or other contra-indications to Coartem® or Malarone® including treatment taken by the volunteer that interferes with Coartem® or Malarone®.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including asplenia.
* Heterozygous or homozygous for sickle cell or homozygous for alpha thalassemia.
* Glucose-6-phosphate dehydrogenase deficiency
* Psychiatric condition that precludes compliance with the protocol; past or present psychoses; disorder requiring lithium; or within five years prior to enrollment, history of suicide plan or attempt.
* Any medical, psychiatric, social condition, or occupational reason that, in the judgment of the investigator, is a contraindication to protocol participation or impairs the volunteer's ability to give informed consent, increases the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* History of 3 or more other immunizations within the six months before administration of the first dose of vaccine.
* Clinically active tuberculosis

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability endpoints | Vaccination to CHMI (or 28 days after last vaccination); CHMI to 28 days after CHMI
  * Solicited local (IV site) and systemic AEs (AEs) observed in the 7 days after each vaccination and each CHMI.
  * Unsolicited AEs observed after the first vaccination until day 28 after the last vaccination for volunteers who do not undergo CHMI#1 (e.g. Group 1, those who do not complete the CHMI portion in Groups 2 and 3, and volunteers in Group 4).
  * Unsolicited AEs observed after the first vaccination until day 28 after the CHMI#1 for volunteers who undergo CHMI#1 3 weeks after the last vaccination (e.g. Groups 2 and 3).
  * Unsolicited AEs observed from day CHMI#2 (which occurs 24 weeks after the last vaccination) until day 28 after CHMI#2 (e.g. Groups 2-5).
Protective Efficacy after CHMI with PfSPZ Challenge (NF54) - CHMI Endpoints | CHMI to 28 days after CHMI
  Number of volunteers that remain parasite negative in each group through day 28 of follow up after CHMI with PfSPZ Challenge (NF54) IV inoculation.
  Three weeks after their last immunization, volunteers in Groups 2 and 3 will under go their first CHMI with 3.2 x 10^3 PfSPZ Challenge (NF54) administered IV. Twenty-four weeks after the last immunization, volunteers from Groups 2 and 3 who underwent the first CHMI and did not become infected will have a second CHMI by IV injection of 3.2x10^3 PfSPZ Challenge (NF54). Volunteers in Groups 4 and 5 will only participate in the second CHMI assessment.
  After CHMI, volunteers will be followed for evidence of infection with blood smears for 28 days.

SECONDARY OUTCOMES:
Immune Responses after PfSPZ Vaccine | 16 months
  Cellular and humoral immune responses will be assessed in the vaccinated volunteers and controls (including central and effector memory responses and breadth and specificity of malaria antibodies).
Protective effect of the high dose PfSPZ Vaccine regimen | CHMI to day 28 after CHMI
  Number of volunteers negative in Group 3 and Group 4 compared to Group 2 through day 28 of follow up after homologous PfSPZ Challenge (NF54) IV inoculation.

OTHER OUTCOMES:
Exploratory Endpoints - Immune Responses | 16 months
  Malaria specific immune responses in Groups 2, 3 and 4 as compared to the malaria naïve volunteers immunized at Vaccine Research Center of the NIH (protocol VRC 312) who received 1.35x10^5 PfSPZ/dose.

CONTACTS AND LOCATIONS:
Overall Officials: Salim Abdulla, MD, PhD, Principal Investigator — Ifakara Health Institute
Locations (1):
- Bagamoyo Research and Training Center, Ifakara Health Institute, Kingani Estate, PO Box 74, Bagamoyo, Tanzania

REFERENCES:
- [Derived] Jongo SA, Shekalaghe SA, Church LWP, Ruben AJ, Schindler T, Zenklusen I, Rutishauser T, Rothen J, Tumbo A, Mkindi C, Mpina M, Mtoro AT, Ishizuka AS, Kassim KR, Milando FA, Qassim M, Juma OA, Mwakasungula S, Simon B, James ER, Abebe Y, Kc N, Chakravarty S, Saverino E, Bakari BM, Billingsley PF, Seder RA, Daubenberger C, Sim BKL, Richie TL, Tanner M, Abdulla S, Hoffman SL. Safety, Immunogenicity, and Protective Efficacy against Controlled Human Malaria Infection of Plasmodium falciparum Sporozoite Vaccine in Tanzanian Adults. Am J Trop Med Hyg. 2018 Aug;99(2):338-349. doi: 10.4269/ajtmh.17-1014. Epub 2018 Jun 21. PMID 29943719
- [Derived] Zenklusen I, Jongo S, Abdulla S, Ramadhani K, Lee Sim BK, Cardamone H, Flannery EL, Nguyen T, Fishbaugher M, Steel RWJ, Betz W, Carmago N, Mikolajczak S, Kappe SHI, Hoffman SL, Sack BK, Daubenberger C. Immunization of Malaria-Preexposed Volunteers With PfSPZ Vaccine Elicits Long-Lived IgM Invasion-Inhibitory and Complement-Fixing Antibodies. J Infect Dis. 2018 Apr 23;217(10):1569-1578. doi: 10.1093/infdis/jiy080. PMID 29438525